CLINICAL TRIAL: NCT04556591
Title: Mobile Technology and Data Analytics to Identify Real-time Predictors of Caregiver Well-Being
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Principal Investigator, Noelle E Carlozzi, Associate Professor of Physical Medicine and Rehabilitation, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: HUM00184455; UL1TR002240 (NIH)
Record Dates: First submitted 2020-09-14; First posted 2020-09-21 (Actual); Results first posted 2023-03-21 (Actual); Last update posted 2023-03-21 (Actual); Status verified 2023-02

CONDITIONS: Caregivers
Keywords: Depression; Insomnia; Stress related disorders; Anxiety
MeSH Terms: conditions — Depression; Sleep Initiation and Maintenance Disorders; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: This behavioral trial will use a two-arm randomized controlled design.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Active Comparator): Participants will wear the Fitbit® and provide daily reports of health related quality of life (HRQOL) over a three-month (90 day) period (without the personalized feedback).
  Interventions: Behavioral: Control
- Just-in-time adaptive intervention (JITAI) (Experimental): Participants will wear the Fitbit®, provide daily reports of health related quality of life (HRQOL) and receive personalized pushes over a three-month (90 day) period.
  Interventions: Behavioral: Just-in-time adaptive intervention (JITAI)

INTERVENTIONS:
Behavioral: Just-in-time adaptive intervention (JITAI) — JITAI is an emerging intervention that incorporates passive mobile sensor data feedback (sleep and activity [step] data from a Fitbit ®), and real-time self-reporting of HRQOL via a study specific app called CareQOL to provide personalized feedback via app alert.
  Arms: Just-in-time adaptive intervention (JITAI)
Behavioral: Control — Participants will wear the Fitbit® and provide daily reports of HRQOL over a three-month (90 day) period
  Arms: Control

SUMMARY:
The purpose of this study is to test whether personalized messages from an easy-to-use mobile app improve mood and stress among care partners and to see if care partners like using the app.

ELIGIBILITY:
Care Partner Inclusion Criteria:

* Provide emotional, physical, and/or financial support/assistance to an individual with spinal cord injury (SCI), Huntington's Disease (HD), or hematopoietic cell transplantation (HCT)
* Have access to necessary resources for participating in a technology-based intervention (smartphone/tablet and internet access) and be willing to use their personal equipment/internet for this study, including downloading the study app and the Fitbit® app on their mobile device
* Care partners of persons with HD: Be caring for an adult (18 years or older) with a clinical diagnosis of HD
* Care partners of persons with SCI: Be caring for an adult (18 years or older) that is ≥1 post-injury and sustained a medically documented SCI at age 16 or older
* Care partners of persons with HCT: Be caring for an adult (18 years or older) who is receiving, has received or is scheduled to receive HCT

Exclusion Criteria:

* Is a professional, paid caregiver (e.g., home health aide)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2020-11-05 (Actual); Primary Completion 2021-06-07 (Actual); Study Completion 2021-06-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Noelle Carlozzi, Ph.D, Principal Investigator — University of Michigan
Locations (1):
- The University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: Yes
Participant data collected during the trial, after de-identification, will be available for sharing with individuals in the scientific community, upon request. The data will be available after the acceptance for publication of the main findings from the final dataset. The University of Michigan Project Manager will coordinate requests for data and maintain documentation for requests and distributions. An institutional data use agreement will be required before data is shared.
Supporting Information: Study Protocol, ICF
Time Frame: The data will be available after the acceptance for publication of the main findings from the final dataset.
Access Criteria: Data is available upon request to the project manager. Requests for data sharing should be emailed to PMR-CODAlab@med.umich.edu.

REFERENCES:
- [Derived] Wang J, Wu Z, Choi SW, Sen S, Yan X, Miner JA, Sander AM, Lyden AK, Troost JP, Carlozzi NE. The Dosing of Mobile-Based Just-in-Time Adaptive Self-Management Prompts for Caregivers: Preliminary Findings From a Pilot Microrandomized Study. JMIR Form Res. 2023 Sep 14;7:e43099. doi: 10.2196/43099. PMID 37707948
- [Derived] Carlozzi NE, Choi SW, Wu Z, Sen S, Troost J, Lyden AK, Miner JA, Graves C, Sander AM. The reliability and validity of the TBI-CareQOL system in four diverse caregiver groups. J Patient Rep Outcomes. 2023 Jun 26;7(1):57. doi: 10.1186/s41687-023-00602-x. PMID 37358716
- [Derived] Carlozzi NE, Choi SW, Wu Z, Troost JP, Lyden AK, Miner JA, Graves CM, Wang J, Yan X, Sen S. An app-based just-in-time-adaptive self-management intervention for care partners: The CareQOL feasibility pilot study. Rehabil Psychol. 2022 Nov;67(4):497-512. doi: 10.1037/rep0000472. PMID 36355640
- [Derived] Carlozzi NE, Choi SW, Wu Z, Miner JA, Lyden AK, Graves C, Wang J, Sen S. An App-Based Just-in-Time Adaptive Self-management Intervention for Care Partners (CareQOL): Protocol for a Pilot Trial. JMIR Res Protoc. 2021 Dec 9;10(12):e32842. doi: 10.2196/32842. PMID 34889775

RESULTS

PARTICIPANT FLOW:
Groups:
- Control: Participants wore the Fitbit® and provided daily reports of health related quality of life (HRQOL) over a three-month (90 day) period (without the personalized feedback).
- Just-in-time Adaptive Intervention (JITAI): Participants wore the Fitbit®, provided daily reports of health related quality of life (HRQOL) and received personalized pushes over a three-month (90 day) period.
  Just-in-time adaptive intervention (JITAI): JITAI is an emerging intervention that incorporates passive mobile sensor data feedback (sleep and activity [step] data from a Fitbit ®), and real-time self-reporting of HRQOL via a study specific app called CareQOL to provide personalized feedback via app alert.
Period: Overall Study
Arm/Group | Control | Just-in-time Adaptive Intervention (JITAI)
Started | 36 | 36
Completed | 33 | 36
Not Completed | 3 | 0
Not completed — Lost to Follow-up | 1 | 0
Not completed — Ineligible after medical record review; documentation for SCI not sufficient | 2 | 0

BASELINE CHARACTERISTICS:
Population: Two persons in the control arm were determined to be ineligible after they were enrolled and completed some study assessments. Both participants were determined to be ineligible by the principal investigator upon medical record review; the medical records did not provide sufficient documentation of spinal cord injury for the persons they cared for. These individuals are included in our summary of adverse events, but they are not included in other reporting as they were deemed ineligible.
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | Just-in-time Adaptive Intervention (JITAI) | Total
Number analyzed (Participants) | 34 | 36 | 70
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.1 (14.5) | 54.4 (13.1) | 55.2 (13.7)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 21 | 28 | 49
  Male | 12 | 8 | 20
  Do not wish to report | 1 | 0 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 2
  Not Hispanic or Latino | 34 | 33 | 67
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 3 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 33 | 29 | 62
  More than one race | 0 | 3 | 3
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 34 | 36 | 70
Caregiver group [Count of Participants; unit: Participants]
  Huntington Disease (HD) | 10 | 11 | 21
  Spinal Cord Injury (SCI) | 9 | 10 | 19
  Hematopoietic cell transplantation (HCT) | 15 | 15 | 30

OUTCOME MEASURES:

1. Primary Outcome: Feasibility and Acceptability as Measured by the Percentage of Agree or Strongly Agree Responses to the Individual Items on the Feasibility Questionnaire
Description: Items are scaled from 1 to 5 to indicate the level of agreement, where "1" indicates "strong disagreement" and "5" indicates "strong agreement".
  Percentages shown are the combined percentage of participants who selected "agree" or "strongly agree" or their equivalent (as labeled).
Time Frame: 3 months of wearing the Fitbit and completing the surveys
Population: one participant did not complete this measure
Measure: Count of Participants; unit: Participants
Groups:
- All Participants, in a Whole Sample: Aggregate data is presented for feasibility and acceptability measures; involvement in the trial is presented for the combined sample as the primary outcome relates to the feasibility and acceptability of the study design rather than the effectiveness of the intervention.
Arm/Group | All Participants, in a Whole Sample
Number analyzed (Participants) | 69
Participants
  Instructions for the Fitbit®️ were easy to understand. | 62
  The Fitbit® was easy to set up. | 63
  The Fitbit® was easy to use. | 64
  The Fitbit® was comfortable to wear. | 60
  The Fitbit® was easy to sync with my phone. | 58
  I was confident using the Fitbit® | 59
  The instructions for the CareQOL app set up were easy to understand. | 66
  The CareQOL app was easy to set up. | 65
  The CareQOL app was easy to use. | 67
  I was confident using the CareQOL app | 67
  I am confident that I was using the CareQOL app correctly. | 65
  The daily questions on the app were easy to understand. | 65
  The daily questions on the app were easy to answer. | 62
  Answering the daily questions fit easily into my routine. | 62
  The number of daily questions to answer on the app was reasonable. | 69
  The monthly surveys on the app were easy to understand. | 66
  The monthly surveys on the app were easy to answer. | 63
  Answering the monthly surveys fit easily into my routine. | 65
  The number of questions in the monthly surveys was reasonable. | 63

2. Secondary Outcome: Attrition as Measured by the Percent of Participants Completing the Study
Time Frame: 3 months of wearing the Fitbit and completing the surveys
Measure: Count of Participants; unit: Participants
Groups:
- All Participants, in a Whole Sample: Aggregate data is presented for feasibility and acceptability measures.
Arm/Group | All Participants, in a Whole Sample
Number analyzed (Participants) | 70
Participants | 69

3. Secondary Outcome: Adherence as Measured by the Percentage of Contributed Data Over the Course of the Study
Description: Contributed data percentages are shown by caregiver group (HD, SCI, HCT) for daily surveys, daily steps, daily sleep, calculated by number of days of data provided divided by number of total possible days that it could be provided.
Time Frame: 3 months of wearing the Fitbit and completing the surveys
Population: Data are presented separately by caregiver group to inform future caregiver studies that may elect to focus on a single caregiver group, as opposed to caregivers more generally.
Measure: Mean (Standard Deviation); unit: percentage of data
Groups:
- HD Care Partners: Data is presented for the HD care partner group for feasibility and acceptability measures.
- SCI Care Partners: Data is presented for the SCI Care Partner group for feasibility and acceptability measures.
- HCT Care Partners: Data is presented for the HCT Care Partner group for feasibility and acceptability measures.
Arm/Group | HD Care Partners | SCI Care Partners | HCT Care Partners
Number analyzed (Participants) | 21 | 19 | 30
percentage of data
  Daily survey | 90 (12) | 84 (14) | 92 (8)
  Daily Steps | 98 (2) | 90 (18) | 99 (2)
  Daily Sleep | 82 (29) | 80 (27) | 90 (21)

ADVERSE EVENTS:
Time Frame: Three months
Description: Two persons in the control arm were determined to be ineligible after they were enrolled. Both participants were determined to be ineligible by the principal investigator upon medical record review; the medical records did not provide sufficient documentation to support a spinal cord injury diagnosis for the persons they cared for. Thus, the data for these two participants is not included since they did not meet study eligibility requirements.
Arm/Group | Control | Just-in-time Adaptive Intervention (JITAI)
All-Cause Mortality (participants affected / at risk) | 0/34 | 0/36
Serious Adverse Events (participants affected / at risk) | 0/34 | 0/36
Other Adverse Events (participants affected / at risk) | 1/34 | 2/36
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control (N=34) | Just-in-time Adaptive Intervention (JITAI) (N=36)
Increased stress (unrelated to study participation) (Social circumstances) | 1 (1) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-04-22): https://cdn.clinicaltrials.gov/large-docs/91/NCT04556591/Prot_SAP_000.pdf
  • Informed Consent Form (2021-02-04): https://cdn.clinicaltrials.gov/large-docs/91/NCT04556591/ICF_001.pdf